CLINICAL TRIAL: NCT05685693
Title: The Effect of ROSA®-Assisted Knee Arthroplasty on Clinical Outcomes
Brief Title: ROSA Knee System vs Conventional Total Knee Arthroplasty
Acronym: ROSA_RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z2021179
Record Dates: First submitted 2022-11-25; First posted 2023-01-17 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Robotic-assisted arthroplasty; Knee arthroplasty; Gait; Metabolic Syndrome; ROSA Knee System; Physical Activity; Cost-effectiveness
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional TKA (Active Comparator): Conventional TKA, with no patient-specific instrumentation or robotic assistance
  Interventions: Procedure: conventional total knee arthroplasty
- Robotic-assisted TKA (Experimental): ROSA Knee System assisted TKA
  Interventions: Procedure: Robotic-assisted total knee arthroplasty (raTKA)

INTERVENTIONS:
Procedure: Robotic-assisted total knee arthroplasty (raTKA) — Robotic-assisted total knee arthroplasty is an orthopaedic surgery that involves replacing the articular surfaces (femoral condyles and tibial plateau) of the knee joint with smooth metal and highly cross-linked polyethylene plastic. The robot (ROSA Knee System, Zimmer Biomet, US) assists in planning and placement of the implants and resection sites.
  Arms: Robotic-assisted TKA
Procedure: conventional total knee arthroplasty — total knee arthroplasty is an orthopaedic surgery that involves replacing the articular surfaces (femoral condyles and tibial plateau) of the knee joint with smooth metal and highly cross-linked polyethylene plastic. In conventional TKAs, no patient-specific instrumentation or robotic assistance is provided.
  Arms: Conventional TKA

SUMMARY:
This is a randomized clinical study, in which 150 patients with end-stage osteoarthritis will be enrolled to ROSA®-assisted knee arthroplasty or conventional knee arthroplasty. Patients are recruited at Zuyderland Medical Center, enrolled pre-operatively and followed up for 12 months post-surgery. In- and exclusion criteria are stated below.

After recruitment, participants will be invited for a pre-operative visit. During this pre-operative visit Informed Consent is signed and completion of patient-reported outcome measures (PROMs) is checked. Additionally, measurements regarding body composition, strength and fitness and metabolic outcomes are performed. Participants will have a blood sample taken. Scans, adverse event and medication use will be confirmed. Participants will receive a ActiGraph for collecting data from physical activity. Of all patients, 72 will undergo additional measurements (gait, proprioception).

During surgery ROSA- and surgery-data will be collected. Post-operative participants will have a 6-weeks, 3-month and 12-month visit. During these visits pre-operative measurements are repeated.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for primary TKA
* age 40-90 years
* Body-Mass-Index 18.5-50.0 kg/m2
* American Society of Anaesthesiologists Class I-III
* Willingness and capability to understand and follow protocol

Exclusion Criteria:

- Rheuma-/trauma-indicated knee arthroplasty

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score | 3-months post-operative
  The Oxford Knee Score (OKS, best to worst 0-48) measures pain intensity and functional limitation of the knee during various activities. The questionnaire consists of 12 items. The maximum total score is 60 and corresponds with the highest pain intensity and functional limitation.
Oxford Knee Score | 12-months post-operative
  The Oxford Knee Score (OKS, best to worst 0-48) measures pain intensity and functional limitation of the knee during various activities. The questionnaire consists of 12 items. The maximum total score is 60 and corresponds with the highest pain intensity and functional limitation.

SECONDARY OUTCOMES:
Quality of Life-Index | Pre-operative, 3-months and 12-months post-operative.
  European Quality of Life-questionnaire-5-dimension-3-level (worst to best, -0.329 to 1.000)
Symptoms | Pre-operative, 3-months and 12-months post-operative.
  Western Ontario and McMaster Universities Osteoarthritis Index (worst to best 0-100)
Pain Catastrophizing | Pre-operative, 3-months and 12-months post-operative.
  Pain Catastrophizing Scale (best to worst, 0-52)
Pain Sensitivity | Pre-operative, 3-months and 12-months post-operative.
  Pain Sensitivity Questionnaire (best to worst, 0-140)
Mobility | Pre-operative, 3-months and 12-months post-operative.
  De Morten Mobility index (worst to best, 0-100)
Complications | During in-patient stay for indicated surgery (up to 5 days)
  Registered complications during hospitalization
Duration of surgery | During surgery
  Registered duration of surgery
Blood loss | During surgery
  Registered blood loss during hospitalization
Length of hospital stay | During in-patient stay for indicated surgery (up to 5 days)
  Duration from patient intake until discharge
Anesthesia | During surgery
  Type of anesthesia used
Stability of the knee | Immediately after the surgery
  Ligament tension, assessed by the ROSA Knee System
Knee implant position | Immediately after the surgery
  Resection, assessed by the ROSA Knee System
Mobility of the knee | During and immediately after the surgery
  Flexion, Extension of knee, assessed by the ROSA Knee System
Mechanical axis of the leg. | 3-months post-surgery
  Hip-Knee-Alignment, by CT
Implant Survival | 90-day and 1-year
  Duration until failure (required revision)
Patient Survival | 90-day and 1-year
  Duration until death
Physical Activity | Pre-operative, 3-months and 12-months post-operative.
  Steps per day, assessed for 7 continuous days using hip-worn accelerometer
Metabolic Syndrome | Pre-operative, 3-months and 12-months post-operative.
  Metabolic Syndrome Severity Scale (no predefined range, higher scores indicate worse outcome)
Body composition | Pre-operative, 3-months and 12-months post-operative.
  Fat mass, measured as % using bioimpedance analysis
Handgrip strength | Pre-operative, 3-months and 12-months post-operative.
  handgrip strength using hand-held dynamometer
Physical condition | Pre-operative, 3-months and 12-months post-operative.
  Completed distance in 2-minute walking
Physical strength | Pre-operative, 3-months and 12-months post-operative.
  Completed sit-to-stand-transfers within 30 seconds
Physical mobility | Pre-operative, 3-months and 12-months post-operative.
  Time to stand up, walk 3m back and forth and sit down again (timed-up-and-go test)
Cost of procedure, implants | During Surgery
  Number implant sizes readily available, and used
Cost of procedure, personnel | During Surgery
  Number of Personnel during surgery
Productivity | Pre-operative, 3-months and 12-months post-operative.
  Institute for Medical Technology Assessment Productivity Cost Questionnaire (worst to best, 0-100)
Medical consumption | Pre-operative, 3-months and 12-months post-operative.
  Institute for Medical Technology Assessment Medical Consumption Questionnaire (outcome in Euro)
Work Ability Index | Pre-operative, 3-months and 12-months post-operative.
  Work Ability Index Questionnaire (worst to best, 0-100)
Work Productivity and Activity Impairment | Pre-operative, 3-months and 12-months post-operative.
  Work Productivity and Activity Impairment-Questionnaire (worst to best, 0-100)

OTHER OUTCOMES:
Gait, walking | Pre-operative, 12-months post-operative
  comfortable walking speed
Gait, sit-to-stand | Pre-operative, 12-months post-operative
  ground reaction force difference between left and right foot during sit-to-stand-transfer
Gait, single-leg-stance | Pre-operative, 12-months post-operative
  standard deviation in center of mass and pressure during single-leg-stance
Proprioception, reaction time | Pre-operative, 12-months post-operative
  Proprioception of the knee will be measured in a motorized carriage. Patients will lay on a hospital bed where their leg is fixed in the motorized carriage. This sled will passively extend and flex the knee. When patients get the sensation of movement, they have to push a button. The reaction time and the angle to sense the movement will be measured digitally.
Proprioception, angle at movement | Pre-operative, 12-months post-operative
  Proprioception of the knee will be measured in a motorized carriage. Patients will lay on a hospital bed where their leg is fixed in the motorized carriage. This sled will passively extend and flex the knee. When patients get the sensation of movement, they have to push a button. The reaction time and the angle to sense the movement will be measured digitally.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Most, PhD, Principal Investigator — Zuyderland Medical Center; Bert Boonen, PhD, Principal Investigator — Zuyderland Medical Center
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eijking HM, Dorling IM, van Haaren EH, Hendrickx R, Nijenhuis T, Schotanus MGM, Bouwman L, Most J, Boonen B. Image-based robotic (ROSA(R) knee system) total knee arthroplasty with inverse kinematic alignment compared to conventional total knee arthroplasty : Study protocol and the inverse kinematic alignment in 8-steps using the ROSA(R) Knee system for knee balancing technique explained. J Orthop Surg Res. 2025 Jan 15;20(1):47. doi: 10.1186/s13018-024-05427-y. PMID 39815282